CLINICAL TRIAL: NCT04905602
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Subcutaneous Administered SHR-1905 in Healthy Subjects and Subjects With Mild Asthma.
Brief Title: A Trial of SHR-1905 in Healthy Subjects and Subjects With Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1905-101
Record Dates: First submitted 2021-05-26; First posted 2021-05-27 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): A single subcutaneous injection of SHR-1905/placebo dose 1 in healthy subjects
  Interventions: Drug: SHR-1905/placebo
- Cohort 2 (Experimental): A single subcutaneous injection of SHR-1905/placebo dose 2 in healthy subjects
  Interventions: Drug: SHR-1905/placebo
- Cohort 3 (Experimental): A single subcutaneous injection of SHR-1905/placebo dose 3 in healthy subjects
  Interventions: Drug: SHR-1905/placebo
- Cohort 4 (Experimental): A single subcutaneous injection of SHR-1905/placebo dose 4 in healthy subjects
  Interventions: Drug: SHR-1905/placebo
- Cohort 5 (Experimental): A single subcutaneous injection of SHR-1905/placebo dose 5 in healthy subjects
  Interventions: Drug: SHR-1905/placebo
- Cohort 6 (Experimental): A single subcutaneous injection of SHR-1905/placebo dose 6 in subjects with mild asthma
  Interventions: Drug: SHR-1905/placebo

INTERVENTIONS:
Drug: SHR-1905/placebo — Drug: SHR-1905 subcutaneous, single dose
  Drug: Placebo subcutaneous, single dose

SUMMARY:
This study is a phase 1 single dose escalation study of SHR-1905 in healthy subjects and subjects with mild asthma. The purpose of the study is to evaluate the safety, tolerability and pharmacokinetics of SHR-1905 in healthy subjects and subjects with mild asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, volunteers to participate in the trial, and provides written informed consent, be able to comply with all the requirements and able to complete the study.
2. Male or female aged between 18 years and 55 years (inclusive) at the date of signed consent form.
3. Total body weight ≥ 45 kg, body mass index (BMI) between 18 and 28 kg/m2 at screening.
4. For healthy subjects, no clinically significant abnormalities in medical history, general physical examination, vital signs, laboratory tests (hematology, urinalysis, blood chemistry, coagulation function and thyroid function) and ECG at the investigator's discretion during screening and baseline.

Exclusion Criteria:

1. Known medical history of severe disease in cardiovascular, liver, kidney, digestive tract, mental, nerve, hematology, metabolic disorders, etc.
2. Severe injuries or major surgeries within 6 months before screening or plan to do surgeries during the trial.
3. Positive hepatitis B virus (HBsAg), hepatitis C virus (HCV-Ab), human immunodeficiency virus (HIV-Ab) at screening.
4. Hyper/Hypotension which define as Systolic blood pressure (SBP) >140mmHg or <90mmHg, or Diastolic blood pressure (DBP)>90mmHg or <40mmHg at screening and at check in.
5. Clinically significant abnormalities in 12-Lead ECG (e.g., For male QTcF > 450msec, for female QTcF > 470msec) at screening and at check in
6. Positive alcohol breath test during baseline visit.
7. Positive nicotine test during screening.
8. Positive urine drug screen during screening.
9. Participation in clinical trials of other investigational drugs or medical devices within 3 months prior to screening or within 5 half-lives of any drugs during screening visit, or in the follow-up period of a clinical study whichever is longer (according to the date of signed consent form) which is defined as have consented and used other investigational drugs (including placebo) or trial medical devices
10. Any other circumstances that, in the investigator's judgment, may increase the risk to the subject, or associated with the subject's participation in and completion of the study or could preclude the evaluation of the subject's response

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
Adverse events | Start of Treatment to end of study (approximately 16 weeks)
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics-AUC0-last | Start of Treatment to end of study (approximately 16 weeks)
  Area under the concentration-time curve from time 0 to last time point after SHR-1905 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to end of study (approximately 16 weeks)
  Area under the concentration-time curve from time 0 to infinity after SHR-1905 administration
Pharmacokinetics-Tmax | Start of Treatment to end of study (approximately 16 weeks)
  Time to Cmax of SHR-1905
Pharmacokinetics-Cmax | Start of Treatment to end of study (approximately 16 weeks)
  Maximum observed concentration of SHR-1905
Pharmacokinetics-CL/F | Start of Treatment to end of study (approximately 16 weeks)
  Apparent clearance of SHR-1905
Pharmacokinetics-V/F | Start of Treament to end of study (approximately 16 weeks)
  Apparent volume of distribution during terminal phase of SHR-1905
Pharmacokinetics-t1/2 | Start of Treatment to end of study (approximately 16 weeks)
  Terminal elimination half-life of SHR-1905
Anti-Drug antibody | Start of Treatment to end of study (approximately 16 weeks)
  The percentage of subjects with positive ADA titers over time for SHR-1905

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China